CLINICAL TRIAL: NCT07281729
Title: Investigation on Risk Factors for Suicide Among Chinese Patients With Mood Disorders
Status: Enrolling by invitation | Type: Observational
Sponsor: Shanghai Mental Health Center (Other)
Responsible Party: Principal Investigator, PENG, Daihui, Chief Physician, Shanghai Mental Health Center
Other Study IDs: 2025-IIT06
Record Dates: First submitted 2025-12-02; First posted 2025-12-15 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Bipolar Disorder；Major Depressive Disorder；Mood Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Main research objective: Through questionnaire surveys, obtain the occurrence levels of self-harm/suicide behaviors, the status of acquired suicidal ability, and their correlations with self-harm/suicide behaviors among patients with mood disorders in mental specialty hospitals and general hospitals.

Main research purpose: (1) Conduct a comprehensive assessment and analysis of the occurrence of suicide/self-harm behaviors, the level of acquired suicidal ability, and their distribution among patients with mood disorders in China; (2) Compare the characteristics and acquired suicidal ability status of patients with mood disorders in mental specialty hospitals and general hospitals' psychological outpatient departments regarding suicide/self-harm behaviors; (3) From multiple dimensions, explore the influencing factors of self-harm/suicide behaviors and acquired suicidal ability in patients with mood disorders, form a list of suicide risk factors and clarify the key risk factors, establish a predictive model for acquired suicidal ability; (4) Through follow-up on whether patients have another occurrence of suicide behavior, clarify the impact of key risk factors on the occurrence of suicide behavior, and verify the effectiveness of the predictive model for acquired suicidal ability.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 16 and 60 years;Presenting at psychiatric hospital or psychological department of general hospital;Willing to cooperate and participate in this study;Informed consent is signed (with additional informed consent provided by guardian for adolescents);Meeting the diagnostic criteria for Mood Disorders as defined by ICD-11.

Exclusion Criteria:

* Inable to comprehend the questionnaire content;Severe organic diseases (e.g., cardiovascular, cerebrovascular, hepatic, or renal impairments) and physically debilitated conditions influencing questionnaire completion;Other situations where participants are unable or unwilling to complete the questionnaire.

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Including people with mood disorders of different ages, genders, occupations, educational levels and cultural backgrounds
Sampling Method: Probability Sample
Enrollment: 25000 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Suicidal behavior/suicide death questionnaire | 1 year
  The one-year follow-up work for 1000 patients (including the main center and 9 representative sub-centers) was completed. Suicidal behavior/suicide death was used as the primary outcome indicator. The follow-up was conducted once every 3 months (via offline interviews; if the patient was unable to come in person, telephone visits were considered), and the content included whether suicidal/self-harming behavior occurred, the current status, and the baseline part of the questionnaire, etc.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Shanghai Mental Health Center, Shanghai, Shanghai Municipality
  - Shanghai Mental Health Center, Shanghai, Xuhui

IPD SHARING:
Plan to Share IPD: No
The prescription data will not be shared with the public. However, if the intervention is effective, the educational materials will be released to the public